CLINICAL TRIAL: NCT05238766
Title: Contextual Behavioral Strategies to Help Parents Adhere to Behavior Plans for Children With Autism
Brief Title: Behavioral Interventions to Increase Parent Adherence With Behavior Plans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Organization for Autism Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00292589
Record Dates: First submitted 2022-01-19; First posted 2022-02-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Family Accommodation; Nonadherence; Behavior Problem
Keywords: Family Accommodation; Nonadherence
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): This arm does not receive any intervention. It will serve as a comparison for the experimental arm.
- Treatment + DEAL (Experimental): Parents in the Treatment plus Defuse Experience Accept Live (T+DEAL) arm will attend five 45-min DEAL sessions with a therapist. Across the five sessions, the therapist will 1) introduce caregivers to behavior change strategies that maximize contact with positive-maintaining contingencies related to adherence, while undermining the contingencies that maintain accommodation, and 2) provide caregivers with new treatment-related committed actions that are sensitive to positive changes in parent-child interactions.
  Interventions: Behavioral: DEAL

INTERVENTIONS:
Behavioral: DEAL — The DEAL protocol is an Acceptance and Commitment Therapy and Behavioral Activation informed clinical protocol to undermine accommodation and help parents adhere with behavioral treatment plan components.
  Arms: Treatment + DEAL

SUMMARY:
Many children with autism demonstrate severe problem behavior (SPB) in the form of self-injury, aggression, and disruptive behavior. Conducting a functional analysis and implementing derived treatments can produce effective behavior plans. Nonetheless, skills training and an effective plan may not be sufficient to produce parent adherence. This applied research proposal describes an approach to target the negative maintaining contingencies supporting parent reinforcement of problem behavior (accommodation) and nonadherence. The intervention, borrowed from Acceptance and Commitment Therapy and Behavioral Activation strategies, is matched specifically to the hypothesized function of the problematic caregiver responses (negative reinforcement). Parents who participate in the proposed investigation will be assigned to either the Defuse Experience Accept Live intervention (DEAL) protocol group or treatment as usual. Five 45-min DEAL sessions will 1) introduce caregivers to behavior change strategies that maximize contact with positive-maintaining contingencies related to adherence, while undermining the contingencies that maintain accommodation, and 2) provide caregivers with new treatment-related committed actions that are sensitive to positive changes in parent-child interactions. Within and between participant analyses will be conducted to determine the effectiveness of the DEAL protocol.

ELIGIBILITY:
Inclusion Criteria:

* Child under the age of 18 years,
* Child is diagnosed with ASD, as confirmed by the Gilliam Autism Rating Scale-3,
* Child problem behavior is socially-maintained as identified via functional analysis,
* Parent is English-speaking, and
* Parent attendance of at least 80% of appointments at entry into the study.

Exclusion Criteria:

* Child is older than 18 years of age,
* Child does not have ASD,
* Child's problem behavior is not socially-maintained,
* Parent does not speak English, and
* Parent attendance at time of study entry is less than 80%.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Accommodation to Adherence Change Score | Change from Time 1 (Week 1) to Time 2 (Week 7)
  Conditional probabilities derived from a contingency space analysis
Experiential Avoidance | Change from Time 1 (Week 1) to Time 2 (Week 7)
  The Acceptance and Action Questionnaire 2nd Edition (AAQ-II) assesses experiential avoidance (EA). The AAQ-II is a 7 item self-report instrument with a range of 7-49. Higher scores are indicative of higher levels of experiential avoidance.
Cognitive Fusion | Change from Time 1 (Week 1) to Time 2 (Week 7)
  The Cognitive Fusion Questionnaire (CFQ) assesses cognitive fusion, or rigidly following self-generated rules. The CFQ is a 7 item self-report instrument with a range of 7-49. Higher scores are indicative of a higher level of cognitive fusion.
Parenting Stress | Change from Time 1 (Week 1) to Time 2 (Week 7)
  The Parenting Stress Index - Short Form (PSI-SF) is a 36 item self-report instrument that measures parenting stress on a 5-point Likert scale. The Parental Distress subscale contains items that resemble statements that a parent might make about their own parenting skills. Self-statements oftentimes may function as rules, which we conceptualize as a more specific measure of parent cognitive fusion. Therefore, we consider high scores on this subscale to be reflective of parent-based cognitive fusion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Kennedy Krieger Institute, Columbia, Maryland

IPD SHARING:
Plan to Share IPD: No
There is not a plan at this time for individual participant data sharing outside of resultant published data. The analytic plan for this trial includes within and between participant analyses. These data may be available at some point in time by specific request.